CLINICAL TRIAL: NCT01055158
Title: Connect: A Pilot Study of Telephone Based Cognitive Behavioral Therapy for HIV Related Depression
Brief Title: Telephone Based Cognitive Behavioral Therapy for HIV Related Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00043648; R34MH080630 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Depression; HIV Infections
Keywords: HIV
MeSH Terms: conditions — Depression; HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone-based CBT (Experimental): A form of CBT delivered over the telephone by a trained, licensed, master's or doctoral level clinician. The intervention consists of approximately 10 sessions conducted over approximately 14 weeks. Each session is approximately 30 to 50 minutes.
  Interventions: Behavioral: Telephone-based CBT
- Control (Active Comparator): Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Telephone-based CBT — A form of CBT delivered over the telephone by a trained, licensed, master's or doctoral level clinician. The intervention consists of approximately 10 sessions conducted over approximately 14 weeks. Each session is approximately 30 to 50 minutes. All sessions begin with a depression rating and agenda setting and end with task assignments and summaries.
  Other Names: CONNECT
  Arms: Telephone-based CBT
Behavioral: Enhanced Usual Care — Participants randomized to this condition will be referred to receive in-person psychotherapy. Research study staff will help participants to set up their first appointment with a psychotherapist.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a telephone-based, cognitive behavioral therapy intervention in the treatment of depression in adults diagnosed with HIV.

DETAILED DESCRIPTION:
Up to 40% of individuals receiving medical care for HIV meet DSM-IV criteria for co-occurring depressive disorder. Individuals with HIV and depressive disorders, compared to those with HIV alone, have been shown to have worse adherence to taking antiretroviral medication, increased HIV related morbidity and among women a higher mortality. Previous research suggests that mental health interventions may lead to improved depressive and HIV related outcomes. However because many HIV infected depressed individuals may have trouble accessing mental health services, there is an urgent need for treatment trials to assess whether treatment of depression targeting patients in urban HIV care settings will result in both improved depressive and HIV related outcomes. The goal of this project is to test the preliminary effectiveness of an adapted telephone-based, cognitive behavioral therapy (CBT) intervention targeting HIV infected depressed individuals receiving care in adult outpatient HIV clinics. A total of 60 HIV infected, depressed individuals receiving care at an urban, outpatient HIV clinic will be randomly assigned to receive either the telephone psychotherapy intervention or enhanced usual care with non-specific telephone contact. The results will provide preliminary data on whether the telephone psychotherapy intervention for HIV infected depressed individuals is effective in reducing depression. The results will also be used to determine feasibility, accessibility, and whether the intervention leads to improved retention and better satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Has a DSM-IV diagnosis of a Depressive Disorder as measured by the mood battery of the MINI
* Has a diagnosis of HIV and is receiving HIV related outpatient care at the Evelyn Jordan Center in Baltimore, MD
* Is able to speak English
* Is able to read English on approximately the 6th grade reading level or higher as measured by the Wide Range Achievement Test 4 (WRAT-4) or by self-report
* Is at least 18 years old
* Has access to a telephone

Exclusion Criteria:

* Meets criteria for dementia by scoring below 10 on the Hopkins HIV Dementia Scale
* Shows signs of serious psychiatric pathology that might either be due to an organic etiology other than HIV, or would generally not be considered treatable solely with psychotherapy, or for whom participation in this protocol might be considered dangerous or unethical
* has a history of serious suicide attempts or is severely suicidal (has ideation, plan, and intent) determined by the MINI
* Patients in psychotherapy are excluded because it is confounded with the study treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | Baseline, Week 8, Week 16
The Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report) (QIDS-SR16) | Baseline, Week 8, Week 16

SECONDARY OUTCOMES:
Provision of Social Relationships (PSR) | Baseline, Week 8, Week 16
Brief COPE | Baseline, Week 8, Week 16
SF-12 Health Survey | Baseline, Week 8, Week 16
Therapist Adherence | Week 1-14
Participant Adherence to Treatment | Week 1-14
Working Alliance Inventory | Week 8, Week 16
Satisfaction Index- Mental Health (SIMH-PW) | Week 8, Week 16
Expectancy Scales | Week 8, Week 16
Adherence to Highly Active Antiretroviral Therapy (HAART) | Baseline, Week 15

CONTACTS AND LOCATIONS:
Overall Officials: Seth S Himelhoch, M.D., M.P.H, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Evelyn Jordan Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Himelhoch S, Medoff D, Maxfield J, Dihmes S, Dixon L, Robinson C, Potts W, Mohr DC. Telephone based cognitive behavioral therapy targeting major depression among urban dwelling, low income people living with HIV/AIDS: results of a randomized controlled trial. AIDS Behav. 2013 Oct;17(8):2756-64. doi: 10.1007/s10461-013-0465-5. PMID 23644816